CLINICAL TRIAL: NCT05673564
Title: Anatomical Resection in Colorectal Liver Metastases Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Other Study IDs: ARCRLM
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: The Characteristics of CRLM Patients Who Would Benefit More From Anatomical Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anatomical resection group: Anatomical resection was defined as resection of 1 or more complete hepatic segments in our study, including bisegmentectomy, right hemihepatectomy, left hemihepatectomy, extended right hemihepatectomy, extended left hemihepatectomy, single segmentectomy, caudate lobectomy, or a combination of these.
  Interventions: Procedure: Anatomical Resection
- nonanatomical resection group: Nonanatomical resection known as wedge resection, was defined as resection of the tumor with a margin of normal parenchyma without regard to hepatic anatomy.

INTERVENTIONS:
Procedure: Anatomical Resection — Based upon the segmental anatomy of the liver according to Couinaud system, AR was defined as resection of 1 or more complete hepatic segments in our study, including bisegmentectomy, right hemihepatectomy, left hemihepatectomy, extended right hemihepatectomy, extended left hemihepatectomy, single segmentectomy, caudate lobectomy, or a combination of these. NAR, known as wedge resection, was defined as resection of the tumor with a margin of normal parenchyma without regard to hepatic anatomy.
  Groups: anatomical resection group

SUMMARY:
The type of liver resection (anatomical resection, AR or nonanatomical resection, NAR) for colorectal liver metastases (CRLM) is subject to debate. The debate may persist because some certain prognostic factors, associated with aggressive biological behavior of tumor, have been overlooked. The aim of our study was to investigate the characteristics of patients who would benefit more from anatomical resection for colorectal liver metastases.

DETAILED DESCRIPTION:
729 patients who underwent hepatic resection of CRLM were retrospectively collected from June 2012and May 2019. Treatment effects between AR and NAR were compared in full subgroup analyses. Tumor relapse-free survival (RFS) was evaluated by a stratified log-rank test and summarized with the use of Kaplan-Meier and Cox proportional hazards methods.

ELIGIBILITY:
Inclusion Criteria:

(1)Age 18-79 years;(2) Histologically proven colorectal adenocarcinoma;

Exclusion Criteria:

(1) the histologic type of tumor was not called adenocarcinoma; (2) peritoneal metastasis; (3) number of liver metastasis >3; (4) simultaneous anatomical and nonanatomical resections; (5) R2 resection; (6) history of previous hepatectomy; (7) incomplete data. The rest of patients were divided into 2 groups: patients undergoing an AR, and patients undergoing a NAR.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was a retrospective cohort study based on our prospectively collected colorectal cancer database. All adult patients who underwent curative-intent liver resection for CRLM between June 2012 and May 2019 at Zhongshan Hospital in Shanghai and had available data on KRAS/NRAS/BRAF status, were eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
RFS | 2012.6.1-2022.6.1
  Relapse-free survival since patients undergoing hepatic resection

SECONDARY OUTCOMES:
OS | 2012.6.1-2022.6.1
  Overall survival since patients undergoing hepatic resection

IPD SHARING:
Plan to Share IPD: No